CLINICAL TRIAL: NCT06851078
Title: Evaluation de l'Administration précoce de lévétiracétam Dans la prévention et le Traitement de l'encéphalopathie au Cours du Choc Septique : Essai randomisé, en Double Aveugle, contrôlé Par Placebo
Brief Title: Evaluation of Early Administration of Levetiracetam in the Prevention and Treatment Encephalopathy in Septic Shock: Randomized, Double-blind, Placebo-controlled Trial
Acronym: KiSS
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: APHP200068
Record Dates: First submitted 2025-02-24; First posted 2025-02-28 (Actual); Last update posted 2025-03-12 (Actual); Status verified 2025-02

CONDITIONS: Septic Shock
MeSH Terms: conditions — Shock, Septic

STUDY DESIGN:
Intervention Model Description: Phase III, multicenter, comparative, randomized, double-blind, placebo-controlled study
Who Masked: Participant, Care Provider, Investigator
Masking Description: Double blind
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Early Levetiracetam administration (Experimental)
  Interventions: Drug: Levetiracetam IV
- Placebo control (Placebo Comparator)
  Interventions: Other: Placebo control

INTERVENTIONS:
Drug: Levetiracetam IV — 1000 mg twice a day during 7 days maximum
  Arms: Early Levetiracetam administration
Other: Placebo control — NaCl 0.9% sodium chloride in the same route and method of administration as experimental treatment
  Arms: Placebo control

SUMMARY:
Sepsis-associated encephalopathy is associated with high mortality rates and long-term neuropsychiatric disorders. Currently, there is no specific treatment for sepsis-associated encephalopathy. Levetiracetam, a broad-spectrum antiepileptic widely used in intensive care units, has neuroprotective properties. We propose the KiSS study, a multicenter, prospective, randomized, double-blind trial with two arms, evaluating the effect of levetiracetam treatment for seven days during septic shock on the occurrence and duration of sepsis-associated encephalopathy.

ELIGIBILITY:
Inclusion criteria :

* Aged 18 years or older
* Hospitalized in intensive care for less than 96 hours
* Presenting with septic shock evolving for less than 24 hours defined by:

  1. Clinically or microbiologically documented infection and
  2. SOFA score ≥ 2 or an increase in SOFA score ≥ 2 points if organ dysfunction was present before the infection and
  3. Need for vasopressor administration to maintain a mean arterial pressure ≥ 65mmHg and
  4. Lactate level > 2mmol/L (18mg/dL) despite adequate fluid resuscitation
* Patient's consent, their next of kin consent, or emergency inclusion

Non inclusion criteria :

* Chronic long-term antiepileptic treatment upon admission or patient with uncontrolled seizures
* Chronic or progressive central neurological pathologies of traumatic, inflammatory, vascular, infectious, neoplastic, or degenerative origin, defined by cognitive impairments preventing independent living or an IQCODE score > 4.5
* Patient with moderate to severe dementia
* Patient with psychiatric history and/or suicide attempts
* Severe head trauma within the past 3 months
* Patients with limitations on active therapies or for whom therapeutic commitment is not maximal
* Patient presenting a prolonged QTc interval on ECG and/or at risk of cardiovascular disease
* Concomitant treatment with Methotrexate during the administration of the investigational treatment
* Allergy to levetiracetam
* Minor patients
* Ongoing pregnancy (blood or urinary βHCG)
* Breastfeeding women
* Patients under guardianship or trusteeship
* Non-affiliation with social security or CMU
* Participation in another interventional trial with a drug that may interact with levetiracetam or may impact the evaluation of KiSS trial outcomes. In case of doubt, please contact the trial's coordinating investigator.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 280 (Estimated)
Dates: Start 2025-03-15 (Estimated); Primary Completion 2027-06-15 (Estimated); Study Completion 2027-06-15 (Estimated)

PRIMARY OUTCOMES:
Number of days alive without delirium or coma | 14 days after randomization

SECONDARY OUTCOMES:
Mortality in intensive care | At day 28
Mortality in intensive care | At day 90
Mortality in hospital | At day 28
Mortality in hospital | At day 90
Overall survival | At day 90
Duration of mechanical ventilation | At day 28
Length of stay in intensive care unit | Up to day 90
Length of stay in hospital | Up to day 90
Occurrence of epileptic seizures | Up to day 14
  From Day 1 to Day 14 (confirmed by EEG or tonic-clonic seizures) and/or occurrence of epileptic abnormalities (periodic epileptic discharges)
Time between cessation of sedation and awakening | At day 90
  Defined by spontaneous eye opening, among patients not deceased under sedation
Severity of cognitive impairment | At day 90
  Evaluated by a telephone survey using Telephone MoCA (Montreal Cognitive Assessment). The scores ranges from 0 to 30.
  A score of 26 or higher is typically considered normal. A score of 25 or lower may indicate cognitive impairment, such as mild cognitive impairment (MCI) or early-stage dementia.
Severity of anxiety and depression | At day 90
  Assessed with HADS (Hospital Anxiety and Depression Scale) scale Score varies from 0 to 21 for each componant (Anxiety and depression) The higher the score, the more severe the anxiety or depression.
Presence of post-traumatic stress (PTSD) | At day 90
  Assessed by IES-R (Impact of Event Scale Revisited) The total score can range from 0 to 88. Higher scores indicate greater trauma-related distress and a higher likelihood of experiencing PTSD symptoms.
Quality of life scoring | At day 90
  Using EQ-5D-5L. It evaluates five dimensions : mobility, self-care, usual activities, pain/discomfort and anxiety/depression and each dimension has five levels : no problems, slight problems, moderate problems, severe problems and extreme problems. Answers are given on a 5-point scale by domain, the higher the score, the poorer the quality of life.
Autonomy in daily life | At day 90
  Using Katz Index of Independence in Activities of Daily Living (ADL) The score varies from 0 to 6, the lower the score, the more dependent the person.

IPD SHARING:
Plan to Share IPD: Undecided